CLINICAL TRIAL: NCT01226368
Title: Epidemiology of Papillomavirus Infection (HPV) on Infected Women by Human Immunodeficience Virus (HIV) in West Indies and French Guiana.
Acronym: HP2V-AG
Status: Completed | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: Fondation de France (Other); Clinique Antilles-Guyane (Other)
Responsible Party: Sponsor
Other Study IDs: 10/B/09
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: 1- Women; 2- HIV Infection; 3- Followed in West Indies and French Guiana for His Infection; 4- Acceptance of the Use of Nadis® Medical Files
Keywords: HIV, HPV, cervical-vaginal smear
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cervix cells
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Biological Sample collection — Cervix cells

SUMMARY:
Cervical cancer is a public health problem. In term of frequency and mortality, it represents in Martinique the third localization the most frequently diagnosed and the fifth cause of death by cancer. Cervical cancer is recognized as viro-inducted. Human papillomavirus (HPV) is the etiologic agent, as a necessary but not sufficient cause, in the cancer genesis. It is estimated than about 70 to 80% of women have been or will be infected with an HPV in their genital life, the risks factors being those of the others sexually transmitted diseases (STD). Most of HPV infection are transient, by spontaneous clearance in a few months of the virus under episomal form.

Carcinogen risk is related to viral persistency which inducts the condition of cellular transformation.

Infection persistency and subsequent carcinogen risk depend of the genotype concerned and of the host immunitary response.

HIV infection is known to be associated with an higher prevalency of one or several infection with HPV-HR.

However, no data about HIV/HPV coinfection prevalency are available nowadays in French overseas department of South America whereas they are the most affected by HIV.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years old or beyond
* Infected with HIV1 or HIV2
* Follow up for HIV infection in one of the center participating in the study and acceptance of the use of Nadis® medical files
* in one of the center participating in the study and acceptance of the use of Nadis® medical files within the context of follow up that should be realized according to the recommandation of undertaking: systematic Pap smear for asymptomatic patient s (expert's report, Pr.P.Yéni) or Pap smear for classical searching of any pathology of the uterine-cervix.
* Acceptance of involvement into the study and collection of non opposition to the realization of HPV search from the sample realized for the Pap smear.

Exclusion Criteria:

* Women under age
* History of total hysterectomy
* Patient not followed for HIV infection in one of the center involved in the study
* Patient that did not accept the use of Nadis® medical files
* Impossibility to realize a Pap smear
* Refusal of study's participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult HIV-Infected women followed in one of the center participating in the study and who has accepted the use of Nadis® medical files.
Sampling Method: Non-Probability Sample
Enrollment: 455 (Actual)
Dates: Start 2010-12; Primary Completion 2011-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Presence of human papillomavirus | 1 day
  Presence of human papillomavirus in women's cervical smear infected with HIV and followed in West Indies and French Guiana

SECONDARY OUTCOMES:
Characterization of Human papillomavirus genotypes | 1 day
  Characterization of Human papillomavirus genotype found in women's cervical smear infected with HIV and followed in West Indies and French Guiana
Presence and the severity of cervical injuries. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie ABEL, MD, Study Director — University Hospital Center of Martinique
Locations (1):
- Centre Hospitalier Universitaire de Fort-de-France, Fort-de-France, Martinique